CLINICAL TRIAL: NCT01169805
Title: Prophylactic Effects of Ondansetron, Ramosetron, and Palonosetron on Patient-Controlled Analgesia Related Nausea and Vomiting After Urologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hae Keum Kil, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2010-0176
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Laparoscopic Marsupialization of Renal Cyst
MeSH Terms: interventions — Ondansetron; ramosetron; Palonosetron

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ONSERAN (Experimental)
  Interventions: Drug: Ondansetron
- NASEA (Experimental)
  Interventions: Drug: Ramosetron
- ALOXI (Experimental)
  Interventions: Drug: Palonosetron
- normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline inj

INTERVENTIONS:
Drug: Ondansetron — Ondansetron/single injection/4 mg/IV
  Other Names: ONSERAN
  Arms: ONSERAN
Drug: Ramosetron — Ramosetron HCl/single injection/0.3mg/IV
  Other Names: NASEA
  Arms: NASEA
Drug: Palonosetron — Palonosetron HCl/single injection/0.075mg/IV
  Other Names: ALOXI
  Arms: ALOXI
Drug: Normal saline inj — normal saline injection 2ml
  Arms: normal saline

SUMMARY:
The aim of this prospective randomized controlled study was to compare the prophylactic effects of intravenous single dose of ondansetron, ramosetron, and palonosetron on PCA-related nausea and vomiting after urologic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Patients aged (20-65 yr) Undergoing Laparoscopic Nephrectomy
* Patients who want a patient-controlled IV analgesia (IV-PCA)

Exclusion Criteria:

* History of allergy or hypersensitivity to 5-HT3 antagonist
* History of severe postoperative nausea/vomiting
* Prolonged QT interval on preoperative EKG
* Hypokalemia, Hypomagnesemia
* Intestinal obstruction
* Pregnant female or breast feeding mother

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
severity of nausea | during 73 hours after surgery
the number of vomiting | during 73 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea